CLINICAL TRIAL: NCT03772899
Title: Fecal Microbial Transplantation in Combination With Immunotherapy in Melanoma Patients (MIMic)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIMic
Record Dates: First submitted 2018-11-16; First posted 2018-12-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Intervention (Experimental): Fecal Microbial Transplantation - all patients registered on study will receive one dose (80-100mg) of FMT. This is a single arm, unblinded study.
  Interventions: Drug: Fecal Microbial Transplantation

INTERVENTIONS:
Drug: Fecal Microbial Transplantation — All patients in this trial will receive FMT at least one week prior to treatment with approved immunotherapy (either pembrolizumab or nivolumab). Samples for FMT are sourced at and by the microbiology group under the supervision of Dr. Silverman at St Joseph's Hospital. Donor screening procedures are described in appendix 4. Transplant will be from one single donor for all participants unless Dr. Silverman's lab considers the need for more than one donor based on availability of donors. There will be no "mixture" of donor samples.
  Donor samples are manufactured into capsules according to Kao et al, 2017.

SUMMARY:
Immunotherapy has helped many cancer patients in the last 5 years by enhancing a patient's immune system to fight cancer. Anti-Programmed Death (PD-1) immunotherapy drugs such as pembrolizumab and nivolumab remove the breaks from cancer-fighting immune cells and have been effective in treating some melanoma patients. Despite the major breakthrough of immunotherapy in oncology treatment, many patients do not respond to this new class of anti-cancer drugs. Recently, evidence suggests that the microorganisms living in a patient's intestines play a major role in modifying the response to anti-PD-1drugs. Patients who respond to these drugs have a unique and healthy group of microorganisms in their gut. Therefore, positive modification of a cancer patient's gut microorganisms to create a more diverse and healthy microbiome may improve the response to immunotherapy. One method of modifying the microbiome is Fecal Microbial Transplantation (FMT) that is already being successfully used in the clinic to treat non-cancer patients with persistent bacterial infections.

In this study, the investigators will combine FMT with the approved immunotherapy drugs pembrolizumab or nivolumab that are the standard of care for the treatment of advanced melanoma. The purpose of this study is to examine the safety of combining these two therapies in melanoma patients. The investigator will use fecal material from a healthy donor selected via our stringent protocol that is Health Canada approved. In addition to assessing the safety of the combination, the investigator will also study the effect of FMT on the immune system and microbial ecosystem of the gut.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18-years old or older
* Patients must have a confirmed diagnosis of unresectable or metastatic cutaneous melanoma (BRAF wild type or mutant)
* Patients with ECOG performance of 0-2
* Patients must be able to provide written informed consent and understand the infectious risks associated with FMT administration
* Must understand non-infectious risks associated with FMT administration
* Ability to ingest capsules
* Understand that data regarding the long-term safety risk of FMT are lacking
* Patients receiving systemic steroids at physiologic doses are permitted to enroll assuming steroid dose is not above the acceptable threshold (> 10 mg prednisone daily or equivalent)
* Have measurable disease as per RECIST version 1.1

Exclusion Criteria:

* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Current or recent [in the last 90 days] exposure to high dose oral or IV corticosteroids

  o Patients who require intermittent use of bronchodilators or local steroid injections are not excluded from the study
* Has a diagnosis of immunodeficiency (e.g. HIV, transplantation) or receiving systemic steroid therapy (>10mg prednisone daily or equivalent) or any other form of immunosuppressive therapy prior to trial treatment
* Ongoing use of antibiotics or previous use of antibiotics in the last two weeks prior to the FMT procedure
* Presence of a chronic intestinal disease (e.g. Celiac, malabsorption, colonic tumor)
* Presence of absolute contra-indications to FMT administration

  * Toxic megacolon
  * Severe dietary allergies (e.g. shellfish, nuts, seafood)
  * Inflammatory bowel disease
  * Anatomic contra-indications to colonoscopy
* Expected to require any other form of systemic or localized anti-neoplastic therapy while on study
* Has a known history of a hematologic malignancy, primary brain tumor or sarcoma, or of another primary solid tumor, unless the patient has undergone potentially curative therapy with no evidence of that disease for five years

  o NOTE: This time requirement also does not apply to patients who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cancers including cervical cancer, breast cancer, melanoma, or other in situ cancers.
* Active central nervous system (CNS) metastases and/or leptomeningeal involvement
* Patients with leptomeningeal disease (leptomeningeal enhancement on MRI/CT imaging and/or positive CSF cytology)
* Has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents.

  o Patients with vitiligo, type I diabetes, resolved childhood asthma/atopy are exceptions to this rule
* A history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has serious concomitant illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders

  o This includes HIV or AIDS-related illness, or active HBV and HCV
* Has an active infection requiring systemic therapy.
* Patient has received a live vaccine within 4 weeks prior to the first dose of treatment

  o Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of combining Fecal Microbial Transplantation (FMT) using intestinal bacteria existing in the stool of healthy donors with immunotherapy in melanoma patients. | 60 months
  Toxicity assessments and concurrent medication review will occur at every visit throughout immunotherapy treatment. Any adverse events after FMT administration will be followed until resolution or until judged stable by the investigator.

SECONDARY OUTCOMES:
Assess Objective Response Rate | At baseline and every 12 weeks thereafter up to 60 months
  To evaluate whether combination of FMT and immunotherapy can enhance antitumor effect in melanoma patients by assessing the objective response rate (ORR; the rate of complete response plus partial response) as per the RECIST 1.1 criteria including immune-related response criteria.
To Evaluate the effect(s) combination FMT and immunotherapy has on the gut microbiome | At baseline, prior to 1st dose of immunotherapy (1 week post FMT) and 2nd dose of immunotherapy (2, 3, or 4 weeks post FMT depending on type of immunotherapy received), and at the 3 month follow-up visit
  Stool sample for microbiome analysis will be collected in the form of used (visibly soiled) toilet paper packed in a labeled biohazard bad and brought with the participant to clinic. The stool sample can be obtained by the patient from a bowel movement up to 3 days prior to the visit.
Evaluate the effect(s) combination FMT and immunotherapy has on changes in immune blood biomarkers | At baseline, prior to 1st dose of immunotherapy (1 week post FMT) and 2nd dose of immunotherapy(2, 3, or 4 weeks post FMT depending on type of immunotherapy received), and at the 3 month follow-up visit
  blood samples will be collected to assess changes in immune blood biomarkers before and after FMT administration by assessing Complete Blood Counts (WBC, HGB, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils)
Evaluate the effect(s) combination FMT and immunotherapy has on changes in immune blood biomarkers | At baseline, prior to 1st dose of immunotherapy (1 week post FMT) and 2nd dose of immunotherapy(2, 3, or 4 weeks post FMT depending on type of immunotherapy received), and at the 3 month follow-up visit
  blood samples will be collected to assess changes in immune blood biomarkers before and after FMT administration by assessing circulating T cells
Evaluate the effect(s) combination FMT and immunotherapy has on changes in immune blood biomarkers | At baseline, prior to 1st dose of immunotherapy (1 week post FMT) and 2nd dose of immunotherapy(2, 3, or 4 weeks post FMT depending on type of immunotherapy received), and at the 3 month follow-up visit
  blood samples will be collected to assess changes in immune blood biomarkers before and after FMT administration by assessing checkpoint molecules including PD-1, PD-L1, TIM-3, LAG-3, TIGIT
Evaluate the effect(s) combination FMT and immunotherapy has on changes in immune blood biomarkers | At baseline, prior to 1st dose of immunotherapy (1 week post FMT) and 2nd dose of immunotherapy(2, 3, or 4 weeks post FMT depending on type of immunotherapy received), and at the 3 month follow-up visit
  blood samples will be collected to assess changes in immune blood biomarkers before and after FMT administration by assessing immune markers such as HLA-DR CD38 and CD28
Evaluate the effect(s) combination FMT and immunotherapy has on patient's metabolomics | At baseline, prior to 1st dose of immunotherapy (1 week post FMT) and 2nd dose of immunotherapy (2, 3, or 4 weeks post FMT depending on type of immunotherapy received), and at the 3 month follow-up visit
  A urine sample will be collected for metabolomics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: John Lenehan, MD, Principal Investigator — London Regional Cancer Program
Locations (3):
- Canada (3):
  - London Regional Cancer Program, London, Ontario
  - CHUM, Montréal, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Routy B, Lenehan JG, Miller WH Jr, Jamal R, Messaoudene M, Daisley BA, Hes C, Al KF, Martinez-Gili L, Puncochar M, Ernst S, Logan D, Belanger K, Esfahani K, Richard C, Ninkov M, Piccinno G, Armanini F, Pinto F, Krishnamoorthy M, Figueredo R, Thebault P, Takis P, Magrill J, Ramsay L, Derosa L, Marchesi JR, Parvathy SN, Elkrief A, Watson IR, Lapointe R, Segata N, Haeryfar SMM, Mullish BH, Silverman MS, Burton JP, Maleki Vareki S. Fecal microbiota transplantation plus anti-PD-1 immunotherapy in advanced melanoma: a phase I trial. Nat Med. 2023 Aug;29(8):2121-2132. doi: 10.1038/s41591-023-02453-x. Epub 2023 Jul 6. PMID 37414899